CLINICAL TRIAL: NCT04143568
Title: Analysis of Circulating Progenitor Cells Levels in Periodontal Disease Patients
Brief Title: Circulating Progenitor Cells Levels in Periodontal Disease Patients
Status: Completed | Type: Observational
Sponsor: University of Messina (Other)
Responsible Party: Principal Investigator, Gaetano Isola, DDS, PhD, Junior Assistant Professor, University of Messina
Other Study IDs: 106-12
Record Dates: First submitted 2019-10-26; First posted 2019-10-29 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Metabolic Disease
MeSH Terms: conditions — Metabolic Diseases | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Evaluation of endothelial progenitor cells level and correlation of endothelial progenitor cells level with periodontal and cardiovascular disease
  Interventions: Other: Observation
- Periodontitis: Evaluation of endothelial progenitor cells level and correlation of endothelial progenitor cells level with periodontal and cardiovascular disease
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Evaluation of endothelial progenitor cells level and correlation of endothelial progenitor cells level with periodontal and cardiovascular disease

SUMMARY:
Recently, a key role played in the ethiology of periodontitis has been highlighted by a subtype of stem cells derived from bone marrow, the circulating endothelial progenitor cells (EPCs). EPCs possess the ability to express surface antigens of endothelial and hematopoietic stem cells and to assist in maintaining vascular integrity and the repair mechanism of the endothelium. Among the main markers for the analysis of EPCs levels are CD34+, CD133+ and the kinase insert domain-containing receptor (KDR). CD34+ and CD133+ originate from hematopoietic stem cell antigens whereas KDR is a specific marker of endothelial cells. More specifically, CD34+ and CD133+/ KDR+ allows less mature and mature EPCs to be evaluated.

DETAILED DESCRIPTION:
The aim of the present study was to investigate the association between endothelial progenitor cells (EPCs) levels subtype (CD133+/KDR+), in patients with periodontitis.

Furthermore, the objective was to determine if the periodontal status influenced CD133+/KDR+ levels.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least 16 teeth
* CP with a minimum of 40% of sites with a clinical attachment level (CAL)

  ≥2mm and probing depth (PD) ≥4mm;
* Presence of at least ≥2 mm of crestal alveolar bone loss verified on digital periapical radiographs
* Presence of ≥40% sites with bleeding on probing (BOP)

Exclusion Criteria:

* Intake of contraceptives

  * Intake of immunosuppressive or anti-inflammatory drugs throughout the last three months prior to the study
  * Status of pregnancy or lactation
  * Previous history of excessive drinking
  * Allergy to local anaesthetic
  * Intake of drugs that may potentially determine gingival hyperplasia such as Hydantoin, Nifedipine, Cyclosporin A or similar drugs.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 79 healthy subjects, 88 patients with CP. Lipid profile and levels of CD133 and C-reactive protein (CRP) were evaluated.
Sampling Method: Non-Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of endothelial progenitor cells level | 1 year
  Changes of endothelial progenitor cells level

CONTACTS AND LOCATIONS:
Locations (1):
- University of Messina, Messina, Italy

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: 5 years
Access Criteria: IRB university of messina